CLINICAL TRIAL: NCT03339245
Title: Effects of Dietary Fructose on Gut Microbiota and Fecal Metabolites in Obese Men and Postmenopausal Women: A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rockefeller University (Other)
Collaborators: Weill Medical College of Cornell University (Other); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: PHO-0956
Record Dates: First submitted 2017-11-07; First posted 2017-11-13 (Actual); Results first posted 2021-03-26 (Actual); Last update posted 2021-03-26 (Actual); Status verified 2021-03

CONDITIONS: Non-Alcoholic Fatty Liver Disease; Obesity
Keywords: obesity; fructose; glucose; fecal microbiota; intestinal permiability; fecal metabolites
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Obesity | interventions — Glucose

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Glucose, Then Fructose (Experimental): Participants first receive Glucose Solution (75 grams) from Day 3 through Day 16 of an inpatient stay with usual diet. After a 2-3 week washout period, they will then receive Fructose Solution (75 Grams) from Day 3 through Day 16 on a second inpatient stay with usual diet.
  Interventions: Other: Fructose Solution (75 Grams); Other: Glucose Solution (75 grams)
- Fructose, Then Glucose (Experimental): Participants first receive Fructose Solution (75 grams) from Day 3 through Day 16 of an inpatient stay with usual diet. After a 2-3 week washout period, they will then receive Glucose Solution (75 grams) from Day 3 through Day 16 on a second inpatient stay with usual diet.
  Interventions: Other: Fructose Solution (75 Grams); Other: Glucose Solution (75 grams)

INTERVENTIONS:
Other: Fructose Solution (75 Grams) — Fructose given in divided doses at breakfast and dinner.
Other: Glucose Solution (75 grams) — Glucose given in divided doses at breakfast and dinner.
  Other Names: Dextrose

SUMMARY:
Non alcoholic fatty liver disease (NAFLD) is the most common cause of abnormal liver function tests in the U.S. (Browning, et al., 2004), ranging from steatosis to end-stage liver disease. Fructose ingestion by the American public has steadily increased since the 1980's, and with it increases in NAFLD, fatty liver hepatitis (NASH), diabetes, obesity, and cardiovascular disease. Foods and beverage in the U.S. are typically sweetened with sucrose (50% glucose and 50% fructose) or high fructose corn syrup (45-58% glucose and 42-55% fructose) (Stanhope, et al., 2009). Research into the role that added fructose plays in the emerging chronic health issues is necessary to affect public policy and provide the connection between fructose and the increasing incidence of these co-morbidities.

There is evidence that gut bacteria contribute to a range of human diseases including those of the liver and gastrointestinal tract. Dietary fructose has been suggested to play a role in the development of these diseases and has been shown to alter gut microbes in animals. If the investigators find that dietary fructose alters bacteria in the human gut, this would suggest a potential targetable link between high fructose diet and disease.

DETAILED DESCRIPTION:
Non- alcoholic fatty liver disease (NAFLD) occurs in 30% of the adult US population (Luther, J., et al., 2015). Eating large amounts of fructose (a dietary sugar) increases liver fat accumulation and worsens NAFLD. In addition, fructose consumption has been shown to greatly increase triglycerides(fat) in the blood after meals, increasing the risk of heart disease,(Stanhope,et al., 2009) insulin resistance and diabetes. Current theories on liver disease caused by consuming fructose focuses on changes in the breakdown of fat by the liver. In experimental animals, fructose feeding changes the bacteria population (microbiota) in the gut, causes NAFLD and NASH, and increases leaking of toxins from the intestine (intestinal permeability) to the blood stream resulting in inflammation.

In humans, fructose consumption rapidly increases liver fat. However, changes in gut microbiota have not been studied. The proposed study will compare the addition of fructose or glucose to the study subjects' usual diet in a crossover design. They will not know which sugar they are receiving.

The Investigators plan to study postmenopausal, moderately obese but healthy women, and moderately obese but healthy men (age 45-70 years) to find out the effect of fructose verses glucose on the bacteria in their stool and inflammation in the bowel. The Investigators hypothesize that adding fructose to the participant's usual diet, compared to glucose, will change stool bacteria composition and the products that the bacteria produce, which may increase intestinal leakage, and increase markers of inflammation in the stool and blood due to this leakage. These changes may contribute to fructose -induced liver disease.

ELIGIBILITY:
Inclusion Criteria:

* Post menopausal female, last menstrual period at least 24 months ago OR male
* Age 45-70
* Willing to consume usual diet with either fructose or glucose added during (2) 16-18 day inpatient stays
* Willing to consume usual diet during 2 week wash-out period at home
* BMI 30.0-39.9
* Willingness not to travel long distances while on study, including wash-out period
* Willingness not to be exposed to new pets while on study including wash-out period

Exclusion Criteria:

* Fasting serum triglycerides >200mg/dl
* Fasting blood glucose >126mg/dl
* Renal function tests >2x Upper limit of normal
* Liver Function Tests > 1.5x Upper limit of normal
* Currently on statins
* Daily use of a cathartic
* Broad spectrum antibiotic use within the past 45 days
* Currently on proton pump inhibitor
* Currently on insulin or oral hypoglycemic agents
* Active viral Hepatitis
* Chronic constipation
* Inflammatory bowel disease
* Chronic diarrhea
* GI resection
* Any evidence of cardiovascular disease on EKG
* History of cardiovascular disease such as coronary artery disease, Coronary Artery Bypass Graft, valve replacement, Myocardial Infarction, stroke / Transient Ischemic attack.
* History of macronutrient malabsorption
* Current smoker. Stopped < 3 months ago.
* Daily alcohol intake equal to 1.5 oz of 40 proof alcohol.
* HIV positive
* Any medical, psychological or social condition that, in the opinion of the Investigator, would jeopardize the health or well-being of the participant during any study procedures or the integrity of the data
* Persons taking probiotics

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2017-12-05 (Actual); Primary Completion 2018-10-02 (Actual); Study Completion 2018-10-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Holt, MD, Principal Investigator — Rockefeller University
Locations (1):
- The Rockefeller University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Browning JD, Szczepaniak LS, Dobbins R, Nuremberg P, Horton JD, Cohen JC, Grundy SM, Hobbs HH. Prevalence of hepatic steatosis in an urban population in the United States: impact of ethnicity. Hepatology. 2004 Dec;40(6):1387-95. doi: 10.1002/hep.20466. PMID 15565570
- [Background] Luther J, Garber JJ, Khalili H, Dave M, Bale SS, Jindal R, Motola DL, Luther S, Bohr S, Jeoung SW, Deshpande V, Singh G, Turner JR, Yarmush ML, Chung RT, Patel SJ. Hepatic Injury in Nonalcoholic Steatohepatitis Contributes to Altered Intestinal Permeability. Cell Mol Gastroenterol Hepatol. 2015 Mar;1(2):222-232. doi: 10.1016/j.jcmgh.2015.01.001. PMID 26405687
- [Background] Stanhope KL, Schwarz JM, Keim NL, Griffen SC, Bremer AA, Graham JL, Hatcher B, Cox CL, Dyachenko A, Zhang W, McGahan JP, Seibert A, Krauss RM, Chiu S, Schaefer EJ, Ai M, Otokozawa S, Nakajima K, Nakano T, Beysen C, Hellerstein MK, Berglund L, Havel PJ. Consuming fructose-sweetened, not glucose-sweetened, beverages increases visceral adiposity and lipids and decreases insulin sensitivity in overweight/obese humans. J Clin Invest. 2009 May;119(5):1322-34. doi: 10.1172/JCI37385. Epub 2009 Apr 20. PMID 19381015
- [Background] Boursier J, Mueller O, Barret M, Machado M, Fizanne L, Araujo-Perez F, Guy CD, Seed PC, Rawls JF, David LA, Hunault G, Oberti F, Cales P, Diehl AM. The severity of nonalcoholic fatty liver disease is associated with gut dysbiosis and shift in the metabolic function of the gut microbiota. Hepatology. 2016 Mar;63(3):764-75. doi: 10.1002/hep.28356. Epub 2016 Jan 13. PMID 26600078

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fructose, Then Glucose | Glucose, Then Fructose
Started | 6 | 7
Completed | 4 (1 withdrawn due to elevated glucose during pre-intervention testing 1 withdrawn for personal reason) | 6 (1 withdrawn due to elevated glucose on baseline testing)
Not Completed | 2 | 1
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: Glucose to Fructose group, 1 was withdrawn due to A/E Total evaluated = 6 Fructose to Glucose group: 1 was withdrawn due to A/E, 1 due to personal reason Total evaluated = 4
Groups:
- Total: Total of all reporting groups
Arm/Group | Glucose, Then Fructose | Fructose, Then Glucose | Total
Number analyzed (Participants) | 7 | 6 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 4 | 10
  >=65 years | 1 | 2 | 3
Age, Continuous [Mean (Full Range); unit: years] — Population: The row population indicates the N in each arm. This is a cross-over study, so each participant received the same intervention but in different order
  years | 58 [50 to 67] | 57 [52 to 65] | 57.6 [50 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 4 | 3 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 6 | 5 | 11
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 4 | 9
  White | 2 | 2 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 6 | 13

OUTCOME MEASURES:

1. Primary Outcome: Difference in the Distribution of Fecal Microbiota in Each Participant
Description: Difference in the distribution of fecal microbiota in each participant, between the fructose versus glucose supplemented diet arms of the study, as measured at the end of each intervention.
Time Frame: assessed at Day 16 of each intervention, up to 64 days
Population: Investigator has retired and access to results for each arm was not available for this outcome. Best efforts were made to obtain the data from the investigator; however, they were unsuccessful.
Arm/Group | Fructose, Then Glucose | Glucose, Then Fructose
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 10 months
Description: Adverse event data are reported per arm/group. Adverse event per intervention are not available because the Investigator has retired. Best efforts were made to obtain and reexamine the adverse event data; however, they were unsuccessful.
Arm/Group | Fructose, Then Glucose | Glucose, Then Fructose
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/6
Other Adverse Events (participants affected / at risk) | 3/4 | 3/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fructose, Then Glucose (N=4) | Glucose, Then Fructose (N=6)
Bloating (Gastrointestinal disorders) | 2 (4) | 3 (3)
nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) — mild nausea resolved spontaneously
elevated blood glucose (Metabolism and nutrition disorders) | 1 (1) | 1 (1) — fasting glucose >125mg/dl
lightheadedness (Nervous system disorders) | 1 (1) | 0 (0) — mild lightheadedness after drinking study sugar, resolved spontaneously
low back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — low back pain after excercising

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-09): https://cdn.clinicaltrials.gov/large-docs/45/NCT03339245/Prot_SAP_000.pdf